CLINICAL TRIAL: NCT00182364
Title: PROphylaxis for ThromboEmbolism in Critical Care Trial (PROTECT Pilot)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 54618366 PROTECT pilot; FGMAEI-0042-048
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Critically Ill; Deep Venous Thrombosis
Keywords: Critically Ill; Deep Venous Thrombosis; Randomized Control Trial; Pilot Study
MeSH Terms: conditions — Critical Illness; Venous Thrombosis | interventions — Dalteparin

INTERVENTIONS:
Drug: Fragmin (Dalteparin) LMWH verus Unfractionated Heparin (UFH)

SUMMARY:
PROTECT Pilot objective is to assess: 1) the feasibility of timely enrollment and complete, blinded study drug administration, 2) the bioaccumulation of LMWH in patients with acquired renal insufficiency and its association with bleeding, 3) the feasibility of scheduled twice weekly lower limb ultrasounds, and 4) recruitment rates for a future randomized trial.

DETAILED DESCRIPTION:
Prophylaxis for Thromboembolism in Critical Care Trial:

PROTECT pilot Study

Background: Critically ill patients have an increased risk of deep venous thrombosis (DVT) due to their acute illness, procedures such as central venous catheterization, and immobility due to sedation and paralysis. Among patients in the intensive care unit (ICU), DVT is an important problem, since thrombus propagation and embolization can lead to potentially fatal pulmonary embolism (PE). Only 1 published randomized trial (n=119) in medical-surgical ICU patients demonstrates that unfractionated heparin (UFH) prevents DVT as compared to no prophylaxis; only 1 published randomized trial (n=223) in mechanically ventilated COPD patients shows that low molecular weight heparin (LMWH) prevents DVT as compared to no prophylaxis. A trial comparing LMWH and UFH for DVT prophylaxis in medical-surgical ICU patients is needed. On one hand, LMWH is likely to be more effective at VTE prevention and is associated with a lower rate of heparin-induced thrombocytopenia (HIT). On the other hand, UFH is likely to be associated with a lower bleeding rate, and is less expensive. The necessity for such a trial is highlighted by the fact that UFH is the dominant method of VTE prophylaxis in critically ill patients in Canada, whereas LMWH is standard of practice in western Europe.

Objectives: The scientific objectives of PROTECT are to determine the effect of LMWH versus UFH on rates of DVT, PE, bleeding, thrombocytopenia and HIT in medical-surgical ICU patients. The feasibility objectives of the PROTECT Pilot are to assess: 1) the feasibility of timely enrollment and complete, blinded study drug administration, 2) the bioaccumulation of LMWH in patients with acquired renal insufficiency and its association with bleeding, 3) the feasibility of scheduled twice weekly lower limb ultrasounds, and 4) recruitment rates for a future randomized trial.

Design: Prospective, concealed, stratified, block randomized, blinded, multicentre trial.

Setting: Canadian medical-surgical university-affiliated ICUs.

Inclusion criteria: Patients >18 years old with an anticipated ICU stay of >72 hours.

Exclusion criteria: Patients admitted to ICU post trauma, orthopedic surgery, cardiac surgery, or neurosurgery, with severe hypertension, DVT, PE or major hemorrhage on admission or within 3 months, coagulopathy, thrombocytopenia, creatinine clearance <30ml/min, or need for therapeutic anticoagulation will be excluded. Patients with documented heparin allergy or HIT, receipt of >2 doses of LMWH or UFH in ICU, contraindication to heparin or blood products, and patients who are pregnant, undergoing withdrawal of life support, or enrolled in a related randomized trial will also be excluded.

Methods: Using centralized telephone randomization, we will allocate 120 patients to dalteparin 5,000 IU daily or unfractionated heparin 5,000 IU twice daily subcutaneously. The ICU team and research personnel will be blinded to study drug. Patients developing creatinine clearance <30 ml/min in ICU will have trough anti-Xa heparin levels; results will be unavailable to the ICU team but used for blinded dose adjustment by the ICU Study Pharmacist. Adherence to study protocol will be maximized using guidelines, interactive education, audit, feedback and reminders. All patients will have bilateral lower limb ultrasound within 48 hours of ICU admission, twice weekly until ICU discharge, upon clinical suspicion of DVT, and within 7 to 10 days after ICU discharge. Patients with a positive or indeterminant ultrasound for proximal DVT will have confirmatory ascending contrast venography if no contraindications exist. We will diagnose PE according to a predefined diagnostic algorithm. We will record bleeding events, thrombocytopenia, HIT and other complications. Patients will be followed throughout their hospital stay. Adjudication Committees blinded to other data will adjudicate indeterminant and positive VTE tests, test complications and bleeding events. We will formally evaluate the success of our feasibility objectives and use intention to treat analysis in this Pilot Study.

Primary Outcome: The primary outcome for the PROTECT Study is objectively confirmed proximal DVT (proven symptomatic or asymptomatic DVT) diagnosed by bilateral lower extremity compression ultrasound, confirmed by venography when possible.

Secondary Outcomes: There are four secondary outcomes: 1) PE diagnosed by the PE Diagnosis algorithm, 2) bleeding, 3) anti-Xa levels associated with heparin dose adjustment, 4) thrombocytopenia and HIT

Relevance: Results of the PROTECT Pilot Study will provide key feasibility and safety data which will serve to plan a larger multicentre trial of LMWH versus UFH for VTE prophylaxis in medical-surgical ICU patients.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to ICU
2. Men and women greater than 18 years of age or older
3. Expected to remain in ICU admission greater than 72 hours

Exclusion Criteria:

1. Contraindications to LMWH or blood products
2. Trauma, post orthopedic surgery, post cardiac surgery or post neurosurgery patients,
3. Uncontrolled hypertension as defined by a systolic blood pressure > 180 mmHg or a diastolic blood pressure > 110 mmHg,
4. Hemorrhagic stroke, DVT, PE or major hemorrhage on admission or within 3 months,
5. Coagulopathy as defined by INR >2 times upper limit of normal [ULN], or PTT >2 times ULN,
6. Renal insufficiency as defined by a creatinine clearance <30ml/min,
7. A need for oral or intravenous or subcutaneous therapeutic anticoagulation,
8. Heparin allergy, proven or suspected heparin-induced thrombocytopenia (HIT),
9. Receipt of >2 doses of UFH or LMWH in ICU,
10. Pregnant or lactating,
11. Withdrawal of life support or limitation of life support,
12. Prior enrollment in this trial
13. Prior enrollment into a related RCT
14. Thrombocytopenia defined platelet count < 100 x 109/L,
15. Bilateral lower limb amputation,
16. Allergy to pork or pork products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-02; Study Completion 2004-02

PRIMARY OUTCOMES:
The primary outcome for the PROTECT Study is objectively confirmed proximal DVT (proven symptomatic or asymptomatic DVT) diagnosed by bilateral lower extremity compression ultrasound, confirmed by venography when possible.

SECONDARY OUTCOMES:
There are four secondary outcomes: 1) PE diagnosed by the PE Diagnosis algorithm, 2) bleeding, 3) anti-Xa levels associated with heparin dose adjustment, 4) thrombocytopenia and HIT

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Cook, MD, Principal Investigator — McMaster University
Locations (16):
- Australia (2):
  - Royal Alfred Hospital, Melbourne
  - Royal North Shore Hospital of Sydney, Sydney
- Canada (14):
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Hamilton Health Science Centre - Hamilton General Hospital, Hamilton, Ontario
  - Hamilton Health Science Centre - McMaster University, Hamilton, Ontario
  - Hamilton Health Science Centre - Henderson Hospital, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Ottawa General Hosptial, Ottawa, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Sunnybrook & Women's College Health Science Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Hopital Sacre Couer, Montreal, Quebec
  - Centre Hospitalier Affilie- Enfant Jesus, Québec, Quebec

REFERENCES:
- [Background] Clarke F, McDonald E, Rocker G, Cook DJ. Research coordinator activities in the ICU: An observational study. Abstract #108. Crit Care Med 2004;31(12)(suppl):A26.
- [Result] Cook DJ, Rocker G, Meade M, Guyatt G, Geerts W, Anderson D, Skrobik Y, Hebert P, Albert M, Cooper J, Bates S, Caco C, Finfer S, Fowler R, Freitag A, Granton J, Jones G, Langevin S, Mehta S, Pagliarello G, Poirier G, Rabbat C, Schiff D, Griffith L, Crowther M; PROTECT Investigators; Canadian Critical Care Trials Group. Prophylaxis of Thromboembolism in Critical Care (PROTECT) Trial: a pilot study. J Crit Care. 2005 Dec;20(4):364-72. doi: 10.1016/j.jcrc.2005.09.010. PMID 16310609
- [Result] McDonald E, Poirier G, Hebert P, Pagliarello J, Rocker G, Langevin S, LeBlanc F F, Mehta S, Skrobik Y, Fowler R, Granton J, Freitag A, Jones G, Cooper DJ, Meade M, Guyatt GH, Anderson D, Geerts W, Crowther M, Zytaruk N, Griffith LE, Cook DJ, for the PROTECT Investigators and Canadian Critical Care Trials Group. PROphylaxis for ThromboEmbolism in Critical care Trial. Blood 2004;104(ii):A1784.
- [Result] Zytaruk N, Cook DJ, Meade M, Rocker G, Poirier G, Langevin S, LeBlanc F, Hebert P, Mehta S, Granton J, Freitag A, Guyatt GH, Anderson D, Geerts W, Crowther M, for the Canadian Critical Care Trials Group. Prophylaxis for thromboembolism in critical care trial: A pilot study. Am J Resp Crit Care Med 2004;169(7):A666.
- [Result] McDonald E, Kho M, Wynne C, Duffet M, McNeil A, Provost L, Rioux A, LaRouche G, Davidson C, McCardle T, Watpool I, Foxall J, Lewis M, Pagliarello J, Jones G, Meade M, Crowther M, Rocker G, Cook DJ, for the Canadian Critical Care Trials Group. Multicenter RCT pilot studies: Exclusion criteria revisited. Am J Resp Crit Care Med 2004;169(7):A257.